CLINICAL TRIAL: NCT03773419
Title: Improving Electronic Written Communication in Persons With Aphasia: A Clinical Trial
Brief Title: Improving Electronic Written Communication in Aphasia
Acronym: T-WRITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: James Madison University (Other)
Responsible Party: Principal Investigator, Leora Cherney, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IFRE17000031
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Aphasia
Keywords: Stroke-related aphasia; Rehabilitation; Writing; Texting
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Texting Intervention (T-WRITE) (Experimental): Computer-based treatment targeting written language via texting (90 minutes a day, 5 days a week for 4 weeks)
  Interventions: Behavioral: Texting Intervention (T-WRITE)
- HandWriting Intervention (ORLA+WTG) (Active Comparator): Computer-based treatment targeting written language via handwriting (90 minutes a day, 5 days a week for 4 weeks)
  Interventions: Behavioral: HandWriting Intervention (ORLA+WTG)

INTERVENTIONS:
Behavioral: Texting Intervention (T-WRITE) — Computer-based intervention, guided by a virtual therapist, that involves repeated listening, reading and writing sentences using a cellular phone
  Arms: Texting Intervention (T-WRITE)
Behavioral: HandWriting Intervention (ORLA+WTG) — Computer-based intervention, guided by a virtual therapist, that involves repeated listening, reading and writing sentences using pen and paper
  Arms: HandWriting Intervention (ORLA+WTG)

SUMMARY:
People with aphasia have difficulty with writing and often struggle to use electronic communication that connects people to one another. The goal of this project is to evaluate the extent to which a novel treatment (T-WRITE) improves written language function and the use of text messaging; we also evaluate whether there are subsequent positive effects on the participant's social connectedness and ultimately health-related quality of life (HRQOL).

T-WRITE involves choral reading and repeated writing of sentences via texting. Participants work intensively and independently at home on a laptop computer. A virtual therapist directs the participant to practice copying and independently writing phrases and short sentences using the typing feature on a cellular phone. The specific objective of this randomized clinical trial is to compare T-WRITE to ORLA+WTG, a similar treatment that targets written expression using handwriting.

DETAILED DESCRIPTION:
An acquired impairment in writing, also known as agraphia, is a characteristic symptom of aphasia, i.e., a language disorder resulting from damage to the language centers of the brain. Written communication via text and instant messaging, electronic mail, and various types of social media has become an increasingly important part of everyday life in our technology driven society. Consequently, difficulty with written expression can significantly restrict people with aphasia from participation in community life, including social, professional, and educational realms. Improving writing in persons with aphasia could improve communication, increase access to information, reduce isolation and facilitate social connectedness. Furthermore, delivering writing treatment via an electronic modality, such as texting, could be particularly advantageous given the increasing reliance on electronic communication. This study investigates the efficacy of T-WRITE, a computer-based writing treatment for aphasia that targets phrase/sentence level writing using texting. Its aims are to: 1) evaluate the efficacy of computer-based texting treatment for improving written communication in persons with aphasia and 2) assess the extent to which improvements in electronic written communication impact social connectedness and health-related quality of life (HRQOL). This will be accomplished via a randomized controlled trial across two sites that compares computer-based texting treatment (T-WRITE) to a control group that receives a hand-writing treatment (ORLA+WTG).

The intervention is delivered via computer using state-of-the-art virtual therapist technology. A perceptive, life-like animated computer agent (virtual therapist), using visible speech, guides the participant so he or she can independently work through the set of choral reading and writing activities (see figure above showing a screen shot of the virtual therapist). The objective is to assure an optimal learning experience in the comfort of the participant's home by using a virtual therapist with accurate visible speech feedback. The virtual therapist reads aloud, speaks with accurate visible speech, highlights and repeats words and sentences, directs the participant to copy/write phrases or sentences, and provides guidance much like a real therapist. The sequence of steps in the ORLA+WTG and the T-WRITE treatments are identical. The output modality for participants randomized to T-WRITE is texting using a cellular phone whereas participants in the ORLA+WTG will hand-write their responses using pen and paper. Participants will practice their writing for 90 minutes a day, 6 days a week for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of an aphasia subsequent to a left-hemisphere infarct(s) that is confirmed by CT scan or MRI
2. Aphasia Quotient score on the Western Aphasia Battery-Revised of 40-85.
3. > 6 months post injury
4. premorbidly right handed, determined by Edinburgh Handedness Inventory
5. completed at least an eighth grade education
6. premorbid proficiency in English by self-report

Exclusion Criteria:

1. any other neurological condition (other than cerebral vascular disease) that could potentially affect cognition or speech, such as Parkinson's Disease, Alzheimer's Dementia, traumatic brain injury.
2. active substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Western Aphasia Battery-Revised (WAB-R) Writing subtest | Change from pre-treatment to post-treatment (i.e. following completion of 36 hours of treatment at 4 weeks)
  Performance-based measure of written language; score ranges from 0 - 100

SECONDARY OUTCOMES:
Stroke and Aphasia Quality of Life Scale (SAQOL-39) | Change from pre-treatment to post-treatment (i.e. following completion of 36 hours of treatment at 4 weeks)
  Self-report measure of health-related quality of life, validated with persons with aphasia; provides a total mean score that ranges from 1 - 39.
The Friendship Scale | Change from pre-treatment to post-treatment (i.e. following completion of 36 hours of treatment at 4 weeks)
  Six-item self-report scale that measures dimensions that contribute to social isolation and social connection. Each item is scored on a 5-point scale (0-4); overall score ranges from 1-24.

CONTACTS AND LOCATIONS:
Overall Officials: Leora Cherney, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (2):
- United States (2):
  - Shirley Ryan AbilityLab, Chicago, Illinois
  - James Madison University, Harrisonburg, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kinsey LE, Lee JB, Larkin EM, Cherney LR. Texting Behaviors of Individuals With Chronic Aphasia: A Descriptive Study. Am J Speech Lang Pathol. 2022 Jan 18;31(1):99-112. doi: 10.1044/2021_AJSLP-20-00287. Epub 2021 Jun 1. PMID 34061572